CLINICAL TRIAL: NCT05761782
Title: Engaging Diverse and Underserved Communities in Cancer Awareness Training and Education (EDUCATE)
Brief Title: Engaging Diverse and Underserved Communities in Cancer Awareness Training and Education
Acronym: EDUCATE
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1992110-1
Record Dates: First submitted 2023-02-16; First posted 2023-03-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer Awareness and Prevention Education
Keywords: Education; Cancer Prevention; Cancer Knowledge; Diverse; Underserved Communities; Cancer Awareness
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University of California, Davis Comprehensive Cancer Center's Catchment Area Population: Behavioral Intervention: Education and Training on Cancer Prevention and Education
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — To educate catchment area residents on modifiable risk factors for cancer (e.g., screening, behavior, vaccination) and the importance of participation in cancer research. Provide participants with educational materials on cancer prevention, screening, and vaccination.

SUMMARY:
The University of California Davis, Comprehensive Cancer Center's (UCDCCC) Office of Community Outreach and Engagement (OCOE) serves the 19 catchment counties which approximately consists of 5 million residents. Currently, the overall catchment population cancer screening rates fall below 80%. The aim of OCOE is to increase cancer education (prevention, screening, and vaccination) and training. Through education, and encouraging participation in routine screening for early detection, this can help increase cancer knowledge. In addition to cancer education, OCOE wants to educate community members regarding modifiable risk factors which include tobacco usage, being overweight/obese (physical inactivity/poor nutrition), and lack of immunizations. By increasing knowledge of cancer prevention, screening, and vaccination this will help community members become more aware of their cancer risk.

DETAILED DESCRIPTION:
Objective: To determine the effects of health education, outreach, and training activities on cancer control and prevention knowledge, attitudes, beliefs, and behaviors among the University of California Davis, Comprehensive Cancer Center's (UCDCCC) catchment area residents. There are 3 Specific Aims for EDUCATE.

Specific Aim 1: To educate catchment area residents on modifiable risk factors for cancer (e.g., screening, behavior, vaccination) and the importance of participation in cancer research.

Specific Aim 2: Provide participants with educational materials on cancer prevention, screening, and vaccination.

Specific Aim 3: Evaluate the effectiveness of the health education, outreach, and training through the analyses of quantitative and qualitative data collected from the health education activities.

ELIGIBILITY:
Inclusion Criteria:

* UCDCCC (University of California, Davis Comprehensive Cancer Center) Catchment Area Population

Exclusion Criteria:

* Above age 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Underserved and Diverse UCDCCC 19-County Catchment Area Population
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
EDUCATE Pre-Presentation Participant Survey | 2 years
  Assessment of participant's experience with cancer screening (Breast, Colorectal, Cervical, Lung or Prostate)
EDUCATE Post-Presentation Participant Survey and Evaluation | 2 years
  Assessment of participant's likelihood to get a cancer screening (Breast, Colorectal, Cervical, Lung or Prostate)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dang, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No